CLINICAL TRIAL: NCT03894956
Title: Special Drug Use-Results Survey of Evaluating Safety and Effectiveness of Humira in Long Term Treatment in Patients With Hidradenitis Suppurativa
Brief Title: Observational Study Evaluating Long-Term Safety and Effectiveness of Humira in Patients With Hidradenitis Suppurativa
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P18-835
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa (HS); Humira; Adalimumab
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants with Hidradenitis Suppurativa (HS): Participants who along with their treating physician have elected for treatment with Humira as per routine clinical practice for the treatment of HS

SUMMARY:
The objective of this study is to evaluate the long-term safety and effectiveness of Humira in patients with Hidradenitis Suppurativa (HS) in real-world clinical practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been prescribed Humira by their treating physician as per routine clinical practice for the treatment of HS.

Exclusion Criteria:

* Participants previously treated with Humira.
* Participants who do not provide consent.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hidradenitis Suppurativa (HS)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who reported any serious infections during the study | Up to Week 52
  Percentage of participants with incidence of serious infections are reported.
Percentage of participants who reported any adverse drug reactions (ADRs) during the study | Up to Week 52
  ADRs will be coded by Medical Dictionary for Regulatory Activities (MedDRA) dictionary.
Percentage of participants who reported any infections during the study | Up to Week 52
  Percentage of participants with incidence of infections are reported.

SECONDARY OUTCOMES:
Percentage of participants achieving "Improved" of overall improvement by physician | Up to Week 52
  Percentage of participants achieving overall improvement (improved, unchanged, impossible to evaluate) is assessed by physician.
Percentage of participants achieving Hidradenitis Suppurativa Clinical Response (HiSCR) | Up to week 52
  HiSCR is defined as at least 50% reduction in the number of abscesses and inflammatory nodules and no increase in abscess count and no increase in draining fistula count relative to baseline.
Change in C-Reactive Protein (CRP) | From Baseline to Week 52
  CRP values are measured as an inflammatory parameter. Low CRP values mean less inflammation.
Change in Patient's global assessment of skin pain | From Baseline to Week 52
  Patient's global assessment of skin pain is evaluated on a 11-point scale with 0 for "no pain" and 10 for "worst skin pain imaginable."
Change in Dermatology Life Quality Index (DLQI) | From Baseline to Week 52
  DLQI is a 10-question validated dermatologic disease questionnaire to measure quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (37):
- Japan (37):
  - Anjou Kousei Hospital /ID# 216741, Anjo-shi, Aichi-ken
  - Ichinomiya Municipal Hospital /ID# 214086, Ichinomiya-shi, Aichi-ken
  - Aichi Medical University Hospital /ID# 215312, Nagakute-shi, Aichi-ken
  - NHO Nagoya Medical Center /ID# 214406, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 214135, Nagoya, Aichi-ken
  - Kimitsu Chuo Hospital /ID# 214733, Kisarazu-shi, Chiba
  - Ehime University Hospital /ID# 214090, Toon-shi, Ehime
  - Kyushu University Hospital /ID# 214092, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan /ID# 214137, Kitakyushu-shi, Fukuoka
  - JA Hiroshima General Hospital /ID# 213472, Hatsukaichi-shi, Hiroshima
  - Sapporo Higashi Tokushukai Hospital /ID# 213865, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 215642, Kobe, Hyōgo
  - Bito Dermatology Clinic /ID# 215316, Kobe, Hyōgo
  - Takarazuka City Hospital /ID# 214088, Takarazuka-shi, Hyōgo
  - Mito Kyodo General Hospital /ID# 214089, Mito, Ibaraki
  - Yokohama City University Medical Center /ID# 216740, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital /ID# 215310, Yokosuka-shi, Kanagawa
  - Kochi Medical School Hospital /ID# 214091, Nankoku-shi, Kochi
  - Kyoto University Hospital /ID# 215315, Kyoto, Kyoto
  - Yokkaichi Municipal Hospital /ID# 215641, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 217830, Sendai, Miyagi
  - Tohoku Rosai Hospital /ID# 214084, Sendai, Miyagi
  - Nara Hospital Kinki University Faculty of Medicine, /ID# 218640, Ikoma-shi, Nara
  - Okayama University Hospital /ID# 215317, Okayama, Okayama-ken
  - University of the Ryukyus Hospital /ID# 214136, Nakagami-gun, Okinawa
  - Kishiwada City Hospital /ID# 213471, Kishiwada-shi, Osaka
  - Kindai University Hospital /ID# 217831, Osakasayama-shi, Osaka
  - Osaka University Hospital /ID# 215314, Suita-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 214087, Takatsuki-shi, Osaka
  - Saitama Medical University Hospital /ID# 215599, Iruma-gun, Saitama
  - Saitama Medical Center /ID# 218639, Kawagoe-shi, Saitama
  - JA Shizuoka Kohseiren Ensh Hospital /ID# 218160, Hamamatsu, Shizuoka
  - Shizuoka City Shizuoka Hospital /ID# 217292, Shizuoka, Shizuoka
  - Toranomon Hospital /ID# 213470, Minato-ku, Tokyo
  - Japan Community Health care Organization Tokyo Yamate Medical Center /ID# 214134, Shinjuku-ku, Tokyo
  - Toyama University Hospital /ID# 214407, Toyama, Toyama
  - Japanese Red Cross Kitami Hospital /ID# 214085, Hokkaido

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hayashi N, Hayama K, Takahashi K, Kurokawa I, Okazaki M, Kashiwagi T, Iwashita E, Terui T. Real-world safety and effectiveness of adalimumab in patients with hidradenitis suppurativa: A 52-week analysis of a postmarketing surveillance study in Japan. J Dermatol. 2023 Aug;50(8):1034-1044. doi: 10.1111/1346-8138.16835. Epub 2023 Jun 2. PMID 37264993
- [Derived] Hayashi N, Hayama K, Takahashi K, Kurokawa I, Okazaki M, Kashiwagi T, Iwashita E, Terui T. Real-world safety and effectiveness of adalimumab in patients with hidradenitis suppurativa: 12-week interim analysis of post-marketing surveillance in Japan. J Dermatol. 2022 Apr;49(4):411-421. doi: 10.1111/1346-8138.16297. Epub 2022 Jan 17. PMID 35040156
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P18-835&Latitude=&Longitude=&LocationName=#additional-resources-section